CLINICAL TRIAL: NCT04662528
Title: A Phase 3, Placebo-Controlled, Randomized, Double-blind, Parallel-arm Trial to Assess the Safety and Efficacy of MAT9001 in Subjects With Severe Hypertriglyceridemia: The AMPLIFY Trial
Brief Title: Safety and Efficacy of MAT9001(Omega-3-pentaenoic Acid) in Subjects With Triglycerides ≥500 mg/dL and <2000 mg/dL
Acronym: AMPLIFY
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: suspended
Sponsor: Matinas Biopharma, Inc (Industry)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MAT-003
Record Dates: First submitted 2020-12-04; First posted 2020-12-10 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Severe Hypertriglyceridemia
MeSH Terms: conditions — Hypertriglyceridemia | interventions — MAT9001

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- MAT9001 (omega-3-pentaenoic acid) (Experimental)
  Interventions: Drug: MAT9001 (omega-3 pentaenoic acid)

INTERVENTIONS:
Drug: Placebo — 4 x 1g capsules/day
  Arms: Placebo
Drug: MAT9001 (omega-3 pentaenoic acid) — 4 x 1g capsules/day
  Arms: MAT9001 (omega-3-pentaenoic acid)

SUMMARY:
To determine the efficacy of MAT9001 compared to placebo in lowering fasting triglyceride levels in subjects with very high fasting triglyceride levels ≥ 500 and < 2000 mg/dL.

DETAILED DESCRIPTION:
This will be a 12-week, randomized, double blind, placebo-controlled safety and efficacy study in men and women ≥18 years of age with fasting triglycerides ≥500 mg/dL and <2000 mg/dL while following a Therapeutic Lifestyle changes (TLC) diet.

ELIGIBILITY:
Inclusion Criteria:

* Fasting triglycerides ≥500 mg/dL and <2000 mg/dL
* Stable lipid-altering drug therapies permitted
* Stable PCSK9 inhibitor use permitted
* BMI ≥20.0 kg/m2
* Willing to maintain a Therapeutic Life Change diet for the duration of the study
* willing to maintain usual physical activity level for the duration of the study
* willing to abstain from alcohol consumption for at least 24 hours prior to each study visit
* agrees not to consume more than 2 meals/week containing fish or seafood
* no plans to change smoking/vaping habits or other nicotine use during the study period
* to be in generally good health on the basis of medical history, physical exam, electrocardiogram (ECG), and screening measurements

Exclusion Criteria:

* Laboratory test result of clinical significance based on the judgment of the Principal Investigator
* A clinically significant GI, endocrine, cardiovascular, renal, hepatic, pulmonary, pancreatic, neurologic, or biliary disorder
* Known lipoprotein lipase impairment or deficiency or Apo C2 deficiency or familial dysbetalipoproteinemia
* Acute or chronic pancreatitis
* Symptomatic gallstone disease (unless previously treated with cholecystectomy).
* Known nephrotic syndrome
* Malabsorption syndrome and/or chronic diarrhea
* Previous bariatric surgery or weight change >3 kg (6.6 lb) during the lead in period.
* Diagnosed hereditary or acquired myopathy
* Uncontrolled diabetes (HbA1c ≥9.5%)
* Uncontrolled hypertension (systolic blood pressure ≥160 mm Hg and/or diastolic blood pressure ≥100 mm Hg)
* Uncontrolled hypothyroidism, thyroid stimulating hormone >5 mIU/L
* History of cancer in the prior 2 years, except non melanoma skin cancer or carcinoma in situ of the cervix
* History of human immunodeficiency virus, hepatitis B, or hepatitis C infection.
* Active systemic infection.
* History of paroxysmal atrial fibrillation, persistent atrial fibrillation, and/or history of ventricular tachycardic arrythmia (e.g., ventricular tachycardia/fibrillation)
* History of a bleeding disorder
* Use of omega 3 drugs /supplements /fortified foods
* Use of bile acid sequestrants, fibrates, or niacin
* Use of dietary supplement(s) that alters lipid metabolism
* Use of weight management drug therapy
* Cardiovascular disease event (myocardial infarction or other acute coronary syndrome, stroke, transient ischemic attack), revascularization procedure
* Female who is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and is unwilling to commit to the use of a medically approved form of contraception throughout the study period
* Known allergy or sensitivity to any ingredients in the study products, including fish, seafood or omega 3 fatty acids
* Been exposed to any investigational drug product within 30 days
* Current or recent history or strong potential for illicit drug or excessive alcohol intake
* A condition that would interfere with ability to provide informed consent or comply with the study protocol, or put the person at undue risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
The percent change from baseline to end of study for MAT9001 versus Placebo | 12 weeks
  Difference between MAT9001 and placebo treatment groups in triglyceride lowering effect

SECONDARY OUTCOMES:
The percent change from baseline to end of study for lipids and lipid biomarkers for MAT9001 versus Placebo | 12 weeks
  Difference between MAT9001 and placebo treatment groups in other lipid and biomarker levels

CONTACTS AND LOCATIONS:
Overall Officials: Judith Johnson, Study Director — Matinas BioPharma

IPD SHARING:
Plan to Share IPD: No